CLINICAL TRIAL: NCT06703216
Title: Pilot Study of Pre-emptive Anakinra for the Prevention of Severe Cytokine Release Syndrome in Children and Young Adults With B-Acute Lymphoblastic Leukemia Receiving Chimeric Antigen Receptor (CAR) T Cells
Brief Title: Pre-emptive Anakinra for Cytokine Event Reduction
Acronym: PACER
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kevin McNerney, Assistant Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-7158; K12TR005104 (NIH)
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: B-Acute Lymphoblastic Leukemia; CAR-T Cell Therapy; Cytokine Release Syndrome; Immune Effector Cell Associated Neurotoxicity Syndrome; Immune Effector Cell Associated Hemophagocytic Lymphohistiocytosis-like Syndrome
Keywords: Anakinra; Cytokine Release Syndrome; CAR-T Therapy; Pediatric; B-acute lymphoblastic leukemia; Prophylaxis; Inflammatory Toxicity; Immune Effector Cell Associated Neurotoxicity Syndrome
MeSH Terms: conditions — Burkitt Lymphoma; Cytokine Release Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Anakinra (Kineret®)

INTERVENTIONS:
Drug: Anakinra (Kineret®) — Pre-emptive Anakinra at the initial onset of CRS.

SUMMARY:
Objectives: The primary objective of this study will be to evaluate the impact of pre-emptive use of anakinra on the rate of severe cytokine release syndrome (CRS) following CD19-directed chimeric antigen receptor (CAR) T-cell therapy for B-acute lymphoblastic leukemia (B-ALL) in children and young adults.

Patient Population: Children and young adults <25 years of age undergoing CAR T-cell therapy for B-ALL with bone marrow disease burden of ≥5% involvement or detectable peripheral blasts within 2 weeks of the initiation of lymphodepleting chemotherapy.

Study Design: This is a pilot single arm study. The investigators will inquire into the efficacy and safety of using anakinra pre-emptively to reduce the rate of severe CRS in patients with >/=5% bone marrow blasts or lymphoblasts in the peripheral blood.

Treatment Plan:

This is a single arm unblinded study in which patients will receive anakinra, 2.5 mg/kg (max 100mg), IV every 12 hours starting at the onset of persistent fever (fever >38.5⁰ C x 2 occurrences separated by at least 4 hours in a 24 hour period). If there is persistence or progression of CRS, anakinra frequency will be increased to 2.5mg/kg IV (max 100mg), every 6 hours. Anakinra will be continued until 48 hours after resolution of CRS and ICANS, and at least 7 days post-CAR T infusion. If dose and frequency of anakinra is increased, the increased dose of anakinra will be continued until 48 hours after resolution of CRS and immune effector cell-associated neurotoxicity syndrome (ICANS) and at least 7 days post-CAR T infusion. For CRS worsening beyond dose escalation of anakinra, CRS will be managed as per standard of care management. Participants will be followed for 12 months following enrollment in the study and disease evaluations will be performed as per routine clinical care following CAR T-cell therapy.

ELIGIBILITY:
• Patient consent and parental assent will be obtained.

NOTE: Signed consent form must be obtained prior to any study procedures. Labs, marrows or other procedures obtained during routine clinical care maybe used for eligibility if obtained within the protocol required windows.

* Patients or their parents/legally authorized representatives (LARs) must have the ability to understand and the willingness to sign a written informed consent document.
* The effects of Anakinra on the developing human fetus are largely unknown. For this reason, patients of child-bearing potential (POCBP) and their partners with sperm-producing reproductive capacity must agree to use adequate contraception from time of informed consent, for the duration of study participation, and for 90 days following completion of Anakinra therapy. Should a POCBP become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. Patients with sperm-producing reproductive capacity (PWSPRC) treated or enrolled on this protocol must also agree to use adequate contraception with partners of childbearing potential from time of informed consent, for the duration of study participation, and 90 days after completion of administration.

Note: A POCBP is any patient (regardless of gender, sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) with an egg-producing reproductive tract who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative serum or urine pregnancy test (women who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
* Patients who are between the age of 1 to 26 years
* Relapsed or refractory B-acute lymphoblastic leukemia

  * 2nd or greater marrow relapse OR
  * Central nervous system (CNS) relapse OR
  * Any relapse after allogeneic hematopoietic stem cell transplant (HSCT) OR
  * Refractory disease defined by not achieving an minimal residual disease (MRD)-negative complete remission (CR) after ≥ 2 chemotherapy cycles (1 cycle for relapsed patients) OR
  * Ineligible for allogeneic HSCT because of:

    * Comorbid disease
    * Other contraindications to allogeneic HSCT conditioning
    * No suitable donor
    * Prior HSCT
    * Declines HSCT as the therapeutic option after documented discussion, with expected outcomes, about the role of HSCT with a HSCT physician
  * Documentation of CD19+ tumor expression in the bone marrow, peripheral blood, cerebrospinal fluid (CSF), or tumor tissue by flow cytometry at relapse, or a recent sample in the case of refractory disease. If the patient has received CD19-directed Pre-emptive anakinra for severe CRS prevention therapy, the flow cytometry should be obtained after this therapy to show CD19 expression.
* Adequate organ function defined as:

  * Alanine aminotransferase (ALT) < 500 U/L
  * Bilirubin ≤2.0 mg/dL
  * Minimum pulmonary reserve defined as ≤Grade 1 dyspnea, pulse oximetry >92% on room air; diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% (corrected for anemia) if pulmonary function tests (PFTs) are clinically appropriate as determined by the treating investigator.
  * Left ventricular shortening fraction ≥ 28% or ejection fraction ≥40% confirmed by echocardiography (ECHO), or adequate ventricular function documented by imaging or a cardiologist.
  * Serum creatinine below the values in the below table, based on age/sex assigned at birth: Maximum Serum Creatinine (mg/dL) Age (years) Male Female 1 to <2 0.6 0.6 2 to <6 0.8 0.8 6 to <10 1.0 1.0 10 to <13 1.2 1.2 13 to <16 1.5 1.4 ≥16 1.7 1.4
* Bone marrow disease burden of ≥5% or peripheral blasts within 2 weeks of the start of lymphodepleting chemotherapy
* Receiving commercially available tisagenlecleucel

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Severe CRS within 30 days of CAR T-cell infusion | 30 days of CAR-T infusion
  The rate of severe CRS, grade ≥3 CRS, as defined by the American Society of Transplantation and Cellular Therapy (ASTCT) consensus guidelines. Participants will have CRS grading each day of hospitalization and every clinical visit within the first 30 days of CAR T-cell infusion.

SECONDARY OUTCOMES:
Complete Remission Rate | 28-35 days post CAR-T infusion
  1. Complete Remission Rate at day 28-35 post-CAR-T
Overall and event-free survival | Up to 12 months post CAR-T infusion
  6- and 12-month overall and event-free survival
CRS and ICANS Severity | Up to 12 months post CAR-T infusion
  Rate and any grade of CRS, any grade ICANS, severe (grade >/=3) ICANS, any grade IEC-HS
Immune effector cell-associated hematotoxicity (ICAHT) Severity | Up to 12 months post CAR-T infusion
  Rate of any grade and grade >/=3 ICAHT as defined by European Hematology Association (EHA)/European Society for Blood and Marrow Transplantation (EBMT) guidelines
Use of tocilizumab or steroids | Within 30 days post CAR T infusion
  Use of tocilizumab and steroids in the treatment of CRS, ICANS, or Immune effector cell-associated hemophagocytic lymphohistiocytosis-like syndrome (IEC-HS)
Infection severity | Within 30 days post CAR T infusion
  Rate of severe infections (as defined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade >/=3)
Inflammatory markers and cell turnover | Within 30 days post CAR T infusion
  Inflammatory markers (C-reactive protein, ferritin) and markers of cell turnover (lactate dehydrogenase and uric acid)
Cell expansion and plasma cytokine profiles | Within 35 days post CAR T infusion
  CAR T-cell expansion and plasma cytokine profiles

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gazeau N, Liang EC, Wu QV, Voutsinas JM, Barba P, Iacoboni G, Kwon M, Ortega JLR, Lopez-Corral L, Hernani R, Ortiz-Maldonado V, Martinez-Cibrian N, Martinez AP, Maziarz RT, Williamson S, Nemecek ER, Shadman M, Cowan AJ, Green DJ, Kimble E, Hirayama AV, Maloney DG, Turtle CJ, Gauthier J. Anakinra for Refractory Cytokine Release Syndrome or Immune Effector Cell-Associated Neurotoxicity Syndrome after Chimeric Antigen Receptor T Cell Therapy. Transplant Cell Ther. 2023 Jul;29(7):430-437. doi: 10.1016/j.jtct.2023.04.001. Epub 2023 Apr 7. PMID 37031746
- [Background] Hines MR, Knight TE, McNerney KO, Leick MB, Jain T, Ahmed S, Frigault MJ, Hill JA, Jain MD, Johnson WT, Lin Y, Mahadeo KM, Maron GM, Marsh RA, Neelapu SS, Nikiforow S, Ombrello AK, Shah NN, Talleur AC, Turicek D, Vatsayan A, Wong SW, Maus MV, Komanduri KV, Berliner N, Henter JI, Perales MA, Frey NV, Teachey DT, Frank MJ, Shah NN. Immune Effector Cell-Associated Hemophagocytic Lymphohistiocytosis-Like Syndrome. Transplant Cell Ther. 2023 Jul;29(7):438.e1-438.e16. doi: 10.1016/j.jtct.2023.03.006. Epub 2023 Mar 9. PMID 36906275
- [Background] Rejeski K, Subklewe M, Aljurf M, Bachy E, Balduzzi A, Barba P, Bruno B, Benjamin R, Carrabba MG, Chabannon C, Ciceri F, Corradini P, Delgado J, Di Blasi R, Greco R, Houot R, Iacoboni G, Jager U, Kersten MJ, Mielke S, Nagler A, Onida F, Peric Z, Roddie C, Ruggeri A, Sanchez-Guijo F, Sanchez-Ortega I, Schneidawind D, Schubert ML, Snowden JA, Thieblemont C, Topp M, Zinzani PL, Gribben JG, Bonini C, Sureda A, Yakoub-Agha I. Immune effector cell-associated hematotoxicity: EHA/EBMT consensus grading and best practice recommendations. Blood. 2023 Sep 7;142(10):865-877. doi: 10.1182/blood.2023020578. PMID 37300386
- [Background] Kineret. Package Insert. Biovitrum AB. December 18th.
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Strati P, Jallouk A, Deng Q, Li X, Feng L, Sun R, Adkins S, Johncy S, Cain T, Steiner RE, Ahmed S, Chihara D, Fayad LE, Iyer SP, Horowitz S, Nastoupil LJ, Nair R, Hassan A, Daoud TE, Hawkins M, Rodriguez MA, Shpall EJ, Ramdial JL, Kebriaei P, Hong DS, Westin JR, Neelapu SS, Green MR. A phase 1 study of prophylactic anakinra to mitigate ICANS in patients with large B-cell lymphoma. Blood Adv. 2023 Nov 14;7(21):6785-6789. doi: 10.1182/bloodadvances.2023010653. No abstract available. PMID 37389847
- [Background] Liang EC, Albittar A, Portuguese AJ, Huang JJ, Wuliji N, Wu Q, De Los Reyes J, Pin N, Torkelson A, Kirchmeier DR. Planned Interim Analysis of a Phase 2 Investigator-Initiated Trial of Anakinra to Prevent CRS and Neurotoxicity after Treatment with Lisocabtagene Maraleucel. Transplantation and Cellular Therapy. 2024;30(2):S179-S80.
- [Background] Frigault MJ, Gallagher KM, Wehrli M, Valles B, Casey K, Lindell K, Trailor M, Cho H, Brown JL, Horick NK. A phase II trial of anakinra for the prevention of CAR-T cell mediated neurotoxicity. Blood. 2021;138:2814.
- [Background] Park JH, Nath K, Devlin SM, Sauter CS, Palomba ML, Shah G, Dahi P, Lin RJ, Scordo M, Perales MA, Shouval R, Tomas AA, Cathcart E, Mead E, Santomasso B, Holodny A, Brentjens RJ, Riviere I, Sadelain M. CD19 CAR T-cell therapy and prophylactic anakinra in relapsed or refractory lymphoma: phase 2 trial interim results. Nat Med. 2023 Jul;29(7):1710-1717. doi: 10.1038/s41591-023-02404-6. Epub 2023 Jul 3. PMID 37400640
- [Background] Hines MR, Keenan C, Maron Alfaro G, Cheng C, Zhou Y, Sharma A, Hurley C, Nichols KE, Gottschalk S, Triplett BM, Talleur AC. Hemophagocytic lymphohistiocytosis-like toxicity (carHLH) after CD19-specific CAR T-cell therapy. Br J Haematol. 2021 Aug;194(4):701-707. doi: 10.1111/bjh.17662. Epub 2021 Jul 15. PMID 34263927
- [Background] Dreyzin A, Jacobsohn D, Angiolillo A, Wistinghausen B, Schore RJ, Perez E, Wells E, Terao J, Bonifant C, Rohatgi R, Dave H, Vatsayan A. Intravenous anakinra for tisagenlecleucel-related toxicities in children and young adults. Pediatr Hematol Oncol. 2022 May;39(4):370-378. doi: 10.1080/08880018.2021.1988012. Epub 2021 Oct 21. No abstract available. PMID 34672243
- [Background] Lichtenstein DA, Schischlik F, Shao L, Steinberg SM, Yates B, Wang HW, Wang Y, Inglefield J, Dulau-Florea A, Ceppi F, Hermida LC, Stringaris K, Dunham K, Homan P, Jailwala P, Mirazee J, Robinson W, Chisholm KM, Yuan C, Stetler-Stevenson M, Ombrello AK, Jin J, Fry TJ, Taylor N, Highfill SL, Jin P, Gardner RA, Shalabi H, Ruppin E, Stroncek DF, Shah NN. Characterization of HLH-like manifestations as a CRS variant in patients receiving CD22 CAR T cells. Blood. 2021 Dec 16;138(24):2469-2484. doi: 10.1182/blood.2021011898. PMID 34525183
- [Background] Diorio C, Vatsayan A, Talleur AC, Annesley C, Jaroscak JJ, Shalabi H, Ombrello AK, Hudspeth M, Maude SL, Gardner RA, Shah NN. Anakinra utilization in refractory pediatric CAR T-cell associated toxicities. Blood Adv. 2022 Jun 14;6(11):3398-3403. doi: 10.1182/bloodadvances.2022006983. No abstract available. PMID 35395068
- [Background] Summerlin J, Wells DA, Anderson MK, Halford Z. A Review of Current and Emerging Therapeutic Options for Hemophagocytic Lymphohistiocytosis. Ann Pharmacother. 2023 Jul;57(7):867-879. doi: 10.1177/10600280221134719. Epub 2022 Nov 9. PMID 36349896
- [Background] Hines MR, von Bahr Greenwood T, Beutel G, Beutel K, Hays JA, Horne A, Janka G, Jordan MB, van Laar JAM, Lachmann G, Lehmberg K, Machowicz R, Miettunen P, La Rosee P, Shakoory B, Zinter MS, Henter JI. Consensus-Based Guidelines for the Recognition, Diagnosis, and Management of Hemophagocytic Lymphohistiocytosis in Critically Ill Children and Adults. Crit Care Med. 2022 May 1;50(5):860-872. doi: 10.1097/CCM.0000000000005361. Epub 2021 Oct 5. PMID 34605776
- [Background] Shakoory B, Carcillo JA, Chatham WW, Amdur RL, Zhao H, Dinarello CA, Cron RQ, Opal SM. Interleukin-1 Receptor Blockade Is Associated With Reduced Mortality in Sepsis Patients With Features of Macrophage Activation Syndrome: Reanalysis of a Prior Phase III Trial. Crit Care Med. 2016 Feb;44(2):275-81. doi: 10.1097/CCM.0000000000001402. PMID 26584195
- [Background] Sonmez HE, Demir S, Bilginer Y, Ozen S. Anakinra treatment in macrophage activation syndrome: a single center experience and systemic review of literature. Clin Rheumatol. 2018 Dec;37(12):3329-3335. doi: 10.1007/s10067-018-4095-1. Epub 2018 Apr 16. PMID 29663156
- [Background] Mehta P, Cron RQ, Hartwell J, Manson JJ, Tattersall RS. Silencing the cytokine storm: the use of intravenous anakinra in haemophagocytic lymphohistiocytosis or macrophage activation syndrome. Lancet Rheumatol. 2020 Jun;2(6):e358-e367. doi: 10.1016/S2665-9913(20)30096-5. Epub 2020 May 4. PMID 32373790
- [Background] Charlesworth JEG, Kavirayani A. Intravenous anakinra for the treatment of haemophagocytic lymphohistiocytosis/macrophage activation syndrome: A systematic review. Eur J Haematol. 2023 Sep;111(3):458-476. doi: 10.1111/ejh.14029. Epub 2023 Jun 21. PMID 37344166
- [Background] Norelli M, Camisa B, Barbiera G, Falcone L, Purevdorj A, Genua M, Sanvito F, Ponzoni M, Doglioni C, Cristofori P, Traversari C, Bordignon C, Ciceri F, Ostuni R, Bonini C, Casucci M, Bondanza A. Monocyte-derived IL-1 and IL-6 are differentially required for cytokine-release syndrome and neurotoxicity due to CAR T cells. Nat Med. 2018 Jun;24(6):739-748. doi: 10.1038/s41591-018-0036-4. Epub 2018 May 28. PMID 29808007
- [Background] Giavridis T, van der Stegen SJC, Eyquem J, Hamieh M, Piersigilli A, Sadelain M. CAR T cell-induced cytokine release syndrome is mediated by macrophages and abated by IL-1 blockade. Nat Med. 2018 Jun;24(6):731-738. doi: 10.1038/s41591-018-0041-7. Epub 2018 May 28. PMID 29808005
- [Background] McNerney KO, Si Lim SJ, Ishikawa K, Dreyzin A, Vatsayan A, Chen JJ, Baggott C, Prabhu S, Pacenta HL, Philips C, Rossoff J, Stefanski HE, Talano JA, Moskop A, Verneris M, Myers D, Karras NA, Brown P, Bonifant CL, Qayed M, Hermiston M, Satwani P, Krupski C, Keating AK, Baumeister SHC, Fabrizio VA, Chinnabhandar V, Egeler E, Mavroukakis S, Curran KJ, Mackall CL, Laetsch TW, Schultz LM. HLH-like toxicities predict poor survival after the use of tisagenlecleucel in children and young adults with B-ALL. Blood Adv. 2023 Jun 27;7(12):2758-2771. doi: 10.1182/bloodadvances.2022008893. PMID 36857419
- [Background] Kadauke S, Myers RM, Li Y, Aplenc R, Baniewicz D, Barrett DM, Barz Leahy A, Callahan C, Dolan JG, Fitzgerald JC, Gladney W, Lacey SF, Liu H, Maude SL, McGuire R, Motley LS, Teachey DT, Wertheim GB, Wray L, DiNofia AM, Grupp SA. Risk-Adapted Preemptive Tocilizumab to Prevent Severe Cytokine Release Syndrome After CTL019 for Pediatric B-Cell Acute Lymphoblastic Leukemia: A Prospective Clinical Trial. J Clin Oncol. 2021 Mar 10;39(8):920-930. doi: 10.1200/JCO.20.02477. Epub 2021 Jan 8. PMID 33417474
- [Background] Schultz LM, Baggott C, Prabhu S, Pacenta HL, Phillips CL, Rossoff J, Stefanski HE, Talano JA, Moskop A, Margossian SP, Verneris MR, Myers GD, Karras NA, Brown PA, Qayed M, Hermiston M, Satwani P, Krupski C, Keating AK, Wilcox R, Rabik CA, Fabrizio VA, Rouce RH, Chinnabhandar V, Kunicki M, Barsan VV, Goksenin AY, Li Y, Mavroukakis S, Egeler E, Curran KJ, Mackall CL, Laetsch TW. Disease Burden Affects Outcomes in Pediatric and Young Adult B-Cell Lymphoblastic Leukemia After Commercial Tisagenlecleucel: A Pediatric Real-World Chimeric Antigen Receptor Consortium Report. J Clin Oncol. 2022 Mar 20;40(9):945-955. doi: 10.1200/JCO.20.03585. Epub 2021 Dec 9. PMID 34882493
- [Background] Pasquini MC, Hu ZH, Curran K, Laetsch T, Locke F, Rouce R, Pulsipher MA, Phillips CL, Keating A, Frigault MJ, Salzberg D, Jaglowski S, Sasine JP, Rosenthal J, Ghosh M, Landsburg D, Margossian S, Martin PL, Kamdar MK, Hematti P, Nikiforow S, Turtle C, Perales MA, Steinert P, Horowitz MM, Moskop A, Pacaud L, Yi L, Chawla R, Bleickardt E, Grupp S. Real-world evidence of tisagenlecleucel for pediatric acute lymphoblastic leukemia and non-Hodgkin lymphoma. Blood Adv. 2020 Nov 10;4(21):5414-5424. doi: 10.1182/bloodadvances.2020003092. PMID 33147337
- [Background] Maude SL, Laetsch TW, Buechner J, Rives S, Boyer M, Bittencourt H, Bader P, Verneris MR, Stefanski HE, Myers GD, Qayed M, De Moerloose B, Hiramatsu H, Schlis K, Davis KL, Martin PL, Nemecek ER, Yanik GA, Peters C, Baruchel A, Boissel N, Mechinaud F, Balduzzi A, Krueger J, June CH, Levine BL, Wood P, Taran T, Leung M, Mueller KT, Zhang Y, Sen K, Lebwohl D, Pulsipher MA, Grupp SA. Tisagenlecleucel in Children and Young Adults with B-Cell Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):439-448. doi: 10.1056/NEJMoa1709866. PMID 29385370